CLINICAL TRIAL: NCT01394315
Title: Diffuse Optical Tomography (DOT) for Monitoring Response to Neoadjuvant (Preoperative) Chemotherapy in Breast Cancer
Acronym: DOT
Status: Terminated | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Yap Yoon Sim, Senior Consultant, National Cancer Centre, Singapore
Other Study IDs: 11-7-BRE
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Breast Neoplasms
Keywords: diffuse optical tomography; response; neoadjuvant chemotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pre-operative biopsy specimens and definitive surgical specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to determine if DOT can detect response early in breast cancer patients undergoing neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The pilot study will enrol up to ten patients over one year. Patients receiving neoadjuvant chemotherapy for breast cancer will undergo baseline clinical examination, mammography, ultrasound, MRI and DOT before commencement of treatment. DOT will be repeated at 1,3,6 weeks after chemotherapy, and at the end of each chemotherapy regimen. Ultrasound will be repeated every 6 weeks and at the end of treatment. Mammography and MRI will be repeated once at the end of treatment before surgery. A breast pathologist will evaluate the subtype of breast cancer and the pathologic response of the operative specimen at the end of treatment. Patient satisfaction questionnaires will be administered to evaluate their preferences for DOT, ultrasound, mammography and MRI scanning at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving neoadjuvant chemotherapy for breast cancer.
* Patients with locally advanced breast tumours or large operable tumours who require neoadjuvant treatment for downstaging.
* Histological confirmation of invasive breast carcinoma.
* Patients with metastatic disease may be eligible if they have oligometastatic disease and breast surgery after neoadjuvant chemotherapy is planned.
* Signed informed consent
* Age equal to or more than 21 years
* Life expectancy greater than 12 weeks.
* ECOG performance status 0-2

Exclusion Criteria:

* Fungating or ulcerated tumours
* Inability to provide informed consent
* Anticipated inability to follow-up patient for response to chemotherapy
* Any contraindication to undergoing ultrasound, MRI, MMG or DOT

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 60 patients are prescribed neaodjuvant chemotherapy for breast cancer at National Cancer Centre Singapore annually. Accrual is expected to be 10 patients per year. Up to 10 patients will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Parameters derived from the optical images acquired with the DOT system | These parameters will be obtained from patients during neoadjuvant chemotherapy process, which is up to an average of 6 months
  The primary parameters derived from the optical images acquired with the DOT system include: The volume of tumor microvasculature V, the total haemoglobin concentration (THC), and the blood volume index BVI (=VC).
  Other available optical parameters are: blood oxygenation in the tumor microvasculature (SO2), its spatial distribution and dynamic fluctuation; dynamic blood perfusion.
  These parameters will be compared with histopathological response.

SECONDARY OUTCOMES:
Change in DOT parameters such as BVI, SO2, blood perfusion dynamic fluctuation | These parameters will be obtained from patients during neoadjuvant chemotherapy process, which is up to an average of 6 months
  The change in DOT parameters such as BVI, SO2, blood perfusion dynamic fluctuation will be correlated with response based on clinical examination, ultrasound, MMG and MRI.
  Standard definitions for clinical response will be used to classify patients into four categories: complete response (CR), partial response (PR), progressive disease (PD) and stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Sim Yap, MBBS, FRACP, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore, Singapore